CLINICAL TRIAL: NCT02148302
Title: A Multi-center Randomized Open-Label Controlled Clinical Trial Evaluating Suction Blister Grafting Utilizing a Novel Harvesting Device (CelluTome©) and Standard of Care vs. Standard of Care Alone in the Treatment of Venous Leg Ulcers
Brief Title: Clinical Trial to Evaluate Blister Graft Utilizing a Novel Harvesting Device for Treatment of Venous Leg Ulcers
Acronym: Cellutome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped by sponsor. No interest in continuing trial due to business changes.
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CELLUTOME-VLU-013
Record Dates: First submitted 2014-01-27; First posted 2014-05-28 (Estimated); Results first posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Impaired Wound Healing; Venous Insufficiency of Leg; Diabetic Ulcers
Keywords: Venous Leg Ulcerations; Epidermal Grafts; Chronic wounds; Clinical trial; Protease levels in chronic wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Harvesting Device (CelluTome©) (Experimental): open-label trial designed to evaluate the safety and effectiveness of Epidermal grafting plus multi-layer compression therapy versus multi-layer compression alone in the healing of venous leg ulcers.
  Epidermal grafting will be applied up to three times in the treatment arm: at day zero, week 4 and week 8.
  A run-in period of two weeks followed by twelve weeks of active treatment
  Interventions: Device: Harvesting Device (CelluTome©)
- Control: SOC alone (No Intervention): The Standard of Care therapy in this study is multi-layer compression therapy. A number of compression bandaging systems are commercially available. The trial will utilize Coban-2 (3M, Minneapolis, MN).

INTERVENTIONS:
Device: Harvesting Device (CelluTome©) — Subjects who continue to meet eligibility criteria will be randomized to one of two groups: (1) Up to 3 applications of Epidermal grafting harvested utilizing the CelluTome® system at day zero, week 4 and week 8, visits plus standard of care (multi-layer compression) (2) Multilayer compression alone.
  Arms: Harvesting Device (CelluTome©)

SUMMARY:
Epidermal grafts are believed to promote healing by two mechanisms: graft take and the promotion of wound healing through the delivery of growth factors and the essential elements of tissue repair and wound healing.28 This study is intended to establish the superior effectiveness of epidermal grafting and multi-layer compression over that of multi-layer compression alone, in the treatment of venous leg ulcers.

Millions of Americans are afflicted with painful, open, draining sores on their lower extremities. These sores are referred to as venous leg ulcerations (VLUs). Under the best of circumstances these ulcers require weeks or months to heal. Not uncommonly wound care specialists see patients who have suffered for years or faced amputation of the limb as their only option to alleviate the pain.

Standard of care will result in healing in 50% of venous leg ulcers in 12 weeks. However, roughly half of patients suffering from venous ulcers will require advanced therapy. Epidermal grafting has been a reconstructive option for decades; however, to date there has not been a reliable and reproducible system to harvest epidermis. The CelluTome® Harvesting System permits the harvesting of epidermal blister grafts at the patient's bedside without the need for anesthesia. The grafts can be easily transferred to the wound bed. In case studies, epidermal grafting appeared to be effective in reducing wound size and accelerating closure of venous leg ulcers.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, controlled open-label study designed to evaluate the safety and effectiveness of epidermal grafting using the CelluTome® system plus multi-layer compression therapy versus multi-layer compression (SOC) in the treatment of venous leg ulcers.

The study will have two phases: Screening and Treatment. The Screening Phase (1 -14 days) is designed to determine whether subjects are eligible to proceed to the Treatment Phase of the study and consists of a series of screening assessments designed to determine eligibility.

At or up to 14 days before the first Screening Phase Visit (S1), written informed consent from the subject will be obtained by the Investigator or suitably qualified designee before the performance of any other protocol-specific procedure.

At the first Screening Phase Visit (S1), the Investigator will select the study (target) ulcer. Each subject will have only one VLU selected as the study (target) ulcer. In the situation where a subject has more than one VLU at the S1 visit, the Investigator will select the largest VLU that meets the eligibility criteria of the protocol as the study (target) ulcer.

Patients whose target ulcer has been treated with compression therapy for the previous two weeks are eligible to enter the treatment phase once all of the inclusion and exclusion criteria are met. If the ulcer has not received compression, the patient should be placed in compression and enrolled in the study after 14 days of compression therapy. Ulcers that have decreased in size by more than 40% during the screening period will be excluded as "rapid healer." Subjects that meet the inclusion/exclusion criteria at the end of screening will be randomized to either the Cellutome graft plus Standard of Care group or just the Standard of Care group. At Treatment Visit 7, subjects in the Standard of Care group that have healed <40% will be allowed to cross over to the Cellutome graft group.

The study will consist of up to 30 centers in the United States each contributing about 10 subjects per center in order to obtain 194 evaluable subjects. The investigators anticipate a 10% drop out rate during the trial therefore a total of 213 subjects will be recruited. This trial employs an adaptive design therefore the enrollment numbers may be reduced or increased based on planned interim analysis.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Adequate arterial flow (Ankle Brachial Pressure Index (ABI) > 0.75. (Calculations will be made using measurements from both posterior tibial and dorsalis pedis arteries as well as both arms), OR Skin Perfusion Pressure (SPP) >30, OR biphasic PVR OR TBI > 0.60 OR TCPO2 > 30mmHg OR adequate perfusion as demonstrated on florescent angiography, LUNA®).
3. Presence of a venous leg ulcer through full skin thickness but not down to muscle, tendon or bone. The largest ulcer will be the index ulcer and the only one included in the study. If other ulcerations are present on the same leg they have to be more than 2 cm apart from the index ulcer.
4. Study ulcer has been present for at least one month prior to the initial screening visit, and is excluded if it has undergone 12 months of continuous high strength compression therapy over its duration.
5. Study ulcer is a minimum of 2.0 cm2 / maximum of 25 cm2 at the randomization visit.
6. The target ulcer has been treated with compression therapy for at least 14 days prior to randomization.
7. Ulcer has a clean, granulating base with minimal adherent slough at the randomization visit.
8. Patient understands / is willing to participate in the clinical study and can comply with weekly visits and follow-up regimen.
9. Patient has read and signed the IRB/IEC approved Informed Consent Form before screening procedures are undertaken.

Exclusion Criteria:

Potential subjects meeting any of the following criteria will be excluded from enrollment and subsequent randomization.

1. Study ulcer(s) deemed by the investigator to be caused by a medical condition other than venous insufficiency. These may include, but are not limited to: fungal ulcerations, malignant ulcerations, and ulcerations due to arterial insufficiency.
2. Study ulcer exhibits clinical signs and symptoms of infection at the SV (screening visit) or TV1 (Treatment Visit 1).
3. Known allergy to the components of the multi-layer compression bandaging, or who cannot tolerate multi-layer compression therapy.
4. Study ulcer is suspicious for cancer should undergo an ulcer biopsy to rule out a carcinoma of the ulcer. The patient may be enrolled after a negative biopsy.
5. Patients with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
6. Study ulcer has been previously treated with tissue engineered materials (e.g. Apligraf® or Dermagraft®) or other scaffold materials (e.g. Oasis, meristem) within the last 30 days
7. Study ulcer requiring negative pressure wound therapy or hyperbaric oxygen during the course of the trial.
8. Ulcers on the dorsum of the foot or with more than 50% of the ulcer below the malleolus are excluded.
9. Pregnant or breast feeding.
10. Known history of having Acquired Immunodeficiency Syndrome (AIDS) or with a history of Human Immunodeficiency Virus (HIV).
11. Known uncontrolled Diabetes Mellitus, as measured by an HbA1c > 10%.
12. Ulcers that have healed more than 40% during the screening phase are excluded.
13. Patients on any investigational drug(s) or therapeutic device(s) within 30 days preceding screening (i.e. S1); or patient or physician anticipates use of any of these therapies by the subject during the course of the study.
14. History of radiation at ulcer site.
15. Presence of one or more medical conditions, including renal, hepatic, hematologic, active auto-immune or immune diseases that, would make the subject an inappropriate candidate for this ulcer healing study.
16. Patients who are unable to understand the aims and objectives of the trial.
17. Presence of any condition(s) which seriously compromises the subject's ability to complete this study, or has a known history of poor adherence with medical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2014-05; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Serena, MD, Principal Investigator — SerenaGroup, Inc.
Locations (18):
- United States (18):
  - Eric Lullove, Dpm, Boca Raton, Florida
  - Advanced Research Institute of Miami, Homestead, Florida
  - Largo Medical Center, Largo, Florida
  - GF Professional Research, Miami Lakes, Florida
  - St Marys Health Care System, Athens, Georgia
  - Michael Miller, Do, Indianapolis, Indiana
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Inspira Health Network, Elmer, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Akron General Medical Center, Akron, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - St John Medical Center, Tulsa, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Summit Health Hospital, Chambersburg, Pennsylvania
  - Saint Vincent Health Center, Erie, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - Regional Medical Center, Orangeburg, South Carolina
  - Pharmakon Medical Research, Harrisonburg, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Harvesting Device (CelluTome©): open-label trial designed to evaluate the safety and effectiveness of Epidermal grafting plus multi-layer compression therapy versus multi-layer compression alone in the healing of venous leg ulcers.
  Epidermal grafting will be applied up to three times in the treatment arm: at day zero, week 4 and week 8.
  A run-in period of two weeks followed by twelve weeks of active treatment
  Harvesting Device (CelluTome©): Subjects who continue to meet eligibility criteria will be randomized to one of two groups: (1) Up to 3 applications of Epidermal grafting harvested utilizing the CelluTome® system at day zero, week 4 and week 8, visits plus standard of care (multi-layer compression) (2) Multilayer compression alone.
Period: Overall Study
Arm/Group | Harvesting Device (CelluTome©) | Control: SOC Alone
Started | 57 | 66
Completed | 57 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Harvesting Device (CelluTome©) | Control: SOC Alone | Total
Number analyzed (Participants) | 57 | 66 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 41 | 78
  >=65 years | 20 | 25 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 37 | 69
  Male | 25 | 29 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 56 | 64 | 120
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 52 | 66 | 118
  Colombia | 5 | 0 | 5
Area at Screening Visit [Mean (Standard Deviation); unit: cm^2] | 8.48 (6.72) | 7.59 (6.81) | 8.04 (6.76)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Healed Wounds
Description: Number of patients experiencing wound healing with epidermal grafting and standard of care vs. standard of care alone
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Harvesting Device (CelluTome©) | Control: SOC Alone
Number analyzed (Participants) | 57 | 66
participants | 11 | 16

2. Secondary Outcome: Wound Area Change at Week 4
Description: Percentage of wound area change at week 4
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of area change
Arm/Group | Harvesting Device (CelluTome©) | Control: SOC Alone
Number analyzed (Participants) | 57 | 66
percentage of area change | 26.8 (20.24) | 27.2 (24.12)

3. Secondary Outcome: Wound Area Change at Week 12
Description: Percentage of wound area change at Week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of area change
Arm/Group | Harvesting Device (CelluTome©) | Control: SOC Alone
Number analyzed (Participants) | 57 | 66
percentage of area change | 41.7 (21) | 47.4 (21.5)

4. Secondary Outcome: Incidence of Adverse Event
Description: Incidence of adverse events with epidermal grafting versus standard of care.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Harvesting Device (CelluTome©) | Control: SOC Alone
Number analyzed (Participants) | 57 | 66
percentage of participants | 28 | 27

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment to subject completion (12 weeks).
Arm/Group | Harvesting Device (CelluTome©) | Control: SOC Alone
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/66
Serious Adverse Events (participants affected / at risk) | 5/57 | 6/66
Other Adverse Events (participants affected / at risk) | 15/57 | 17/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Harvesting Device (CelluTome©) (N=57) | Control: SOC Alone (N=66)
Infection (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6) — Infection of venous leg ulcer
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Harvesting Device (CelluTome©) (N=57) | Control: SOC Alone (N=66)
Cold (General disorders) | 15 (15) | 17 (17)

LIMITATIONS AND CAVEATS:
The study was terminated before protocol enrollment could be reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT02148302/Prot_SAP_000.pdf